CLINICAL TRIAL: NCT01933737
Title: Kinesio Taping Effect on Postural Balance in Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The collected data was finished
Sponsor: University of Franca (Other)
Responsible Party: Principal Investigator, Paulo Roberto Veiga Quemelo, Paulo Quemelo, University of Franca
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNIFRAN
Record Dates: First submitted 2013-08-21; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Accidental Falls
Keywords: postural balance;; elderly;; proprioception;; prevention;; fall

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio Taping Group (Experimental): The Kinesio Taping group (KTG) (n = 31 elderly women) were submitted to the protocol of applying Kinesio Taping for gastrocnemius muscle and the muscles of the median foot. The application of the tapes was bilateral limbs. The subjects were evaluated post-application and 48 hours after application of the tape.
  Interventions: Device: Kinesio Taping
- Placebo tape group (Experimental): The placebo tape group (PTG) (n = 31 elderly women) were submitted to the protocol of applying placebo tape (3M Micropore) for gastrocnemius muscle and the muscles of the median foot in the same way that KTG. The application of the tapes was bilateral limbs. The subjects were evaluated post-application and 48 hours after application of the tape.
  Interventions: Device: 3M Micropore

INTERVENTIONS:
Device: Kinesio Taping — The Kinesio Taping group (KTG) (n = 31 elderly women) were submitted to the protocol of applying Kinesio Taping for gastrocnemius muscle and the muscles of the median foot. The application of the tapes was bilateral limbs. The subjects were evaluated post-application and 48 hours after application of the tape.
  Arms: Kinesio Taping Group
Device: 3M Micropore — The placebo tape group (PTG) (n = 31 elderly women) were submitted to the protocol of applying placebo tape (3M Micropore) for gastrocnemius muscle and the muscles of the median foot in the same way that KTG. The application of the tapes was bilateral limbs. The subjects were evaluated post-application and 48 hours after application of the tape.
  Arms: Placebo tape group

SUMMARY:
The elderly population has increased significantly in the last years. The number of falls has also increased due to the decrease of balance. The Kinesio Taping (KT) is a method with the aim to improve muscle physiology, proprioception, coordination and balance. The aim of the study was to investigate the effect of KT on postural balance in the elderly. We evaluated 62 elderly with a mean age of 67.98±5.321, female, submitted to the protocol for the application of KT in gastrocnemius muscles of the midfoot and a placebo tape (3M Micropore) in the control group. The application of the tapes was bilateral. Half of the participants (n=31) received KT in the lower limbs, while the control group (n=31) was applied placebo tape. To analysis of posture and balance, we used a force plate to record stabilometric signals. Both groups were evaluated post-application and 48 hours after application of the tape. The variables used were total displacement in centimeters (cm), amplitude AP (anterior-posterior) and ML (medial-lateral) in centimeters, area (cm²) and speed AP and ML in centimeters for seconds. The experimental protocol was performed in standing posture and the subjects were instructed to stand with feet apart, eyes open to look at the fixed point 1.5 m from force plate in a horizontal direction. It was requested that the elderly maintain the position for a time of 40 seconds to collect data The data were collected immediately post application of tapes and after 48 hours. The data was tabulated, descriptive statistics were calculated. Statistical analysis was performed using the GraphPad Prism 4.0 software (Prism, Chicago, IL). The Kolmogorov Smirnov test was used to verify the data distribution. Differences between the means were evaluated using the Student T test for the normally distributed data, and using the Mann-Whitney test for the data not normally distributed. Significance levels were set at p<0.05.

DETAILED DESCRIPTION:
The Kinesio Taping Group (KTG) was composed of 31 participants that received the application of KT (K-Taping®) on the gastrocnemius muscle and the muscles of the midfoot. The placebo tape group (PTG) was composed of 31 participants that received the application of a placebo tape (3M Micropore®) on the same muscles of both limbs. The order of application of KT tape and placebo was conducted randomly among the elderly. Before the tape applying the site was cleaned with 70% ethanol for better fixation of the tape and for both groups were determined the application technique in "I" shaped. This technique consist in placing two tapes that format. The first tape was placed along the length of the plantar aponeurosis fixed point in the middle third of the medial gastrocnemius muscle to the metatarsal phalangeal joint. The second tape was also applied in "I" shaped without fixed point was placed around the midfoot arch in the direction of tension lines to assist with the metatarsal arch support.

ELIGIBILITY:
Inclusion Criteria:

* elderly, gender female

Exclusion Criteria:

* No severe orthopedic diseases

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Force plate to postural balance | 6 months
  To analysis of posture and balance, we used a force plate to record stabilometric signals. Both groups were evaluated post-application and 48 hours after application of the tape. The variables used were total displacement in centimeters (cm), amplitude AP (anterior-posterior) and ML (medial-lateral) in centimeters, area (cm²) and speed AP and ML in centimeters for seconds. We did not observe adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RV Quemelo, PhD, Principal Investigator — University of Franca
Locations (1):
- University of Franca, Franca, São Paulo, Brazil

REFERENCES:
- [Result] Lins CA, Neto FL, Amorim AB, Macedo Lde B, Brasileiro JS. Kinesio Taping((R)) does not alter neuromuscular performance of femoral quadriceps or lower limb function in healthy subjects: randomized, blind, controlled, clinical trial. Man Ther. 2013 Feb;18(1):41-5. doi: 10.1016/j.math.2012.06.009. Epub 2012 Jul 15. PMID 22796389